CLINICAL TRIAL: NCT06300554
Title: 10th Mountain Healthy Minds Program App Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-1653; A171600 (Other: UW Madison); Version 1/26/2024 (Other: UW Madison)
Record Dates: First submitted 2024-02-21; First posted 2024-03-08 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Well-Being, Psychological
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants from the 10th Mountain Division (Experimental)
  Interventions: Device: Healthy Minds Program App

INTERVENTIONS:
Device: Healthy Minds Program App — freely available well-being app

SUMMARY:
The purpose of the study is to evaluate the acceptability, feasibility, and preliminary effects of the Healthy Minds Program (HMP) App in approximately 150 active duty military members.

DETAILED DESCRIPTION:
Participants will be informed about the study during regularly scheduled activities. They will be informed that enrolling in the study is voluntary.

Participants will complete a 10-15 minute battery of questionnaires at baseline and post-test. In between these assessments, they will be asked to download and use the Healthy Minds Program app for 4 weeks. Post-test assessment will occur following the 4-week intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Active duty military at the 10th Mountain Division

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-22 (Actual); Study Completion 2024-10-22 (Actual)

PRIMARY OUTCOMES:
System Usability Scale Score | post-test (up to 4 weeks)
  Scored from 1 to 5 where higher scores indicate increased usability.
Acceptability of Intervention Measure (AIM) | post-test (up to 4 weeks)
  Scored from 1 to 5 where higher scores indicate increased acceptability.
Intervention Appropriateness Measure (IAM) | post-test (up to 4 weeks)
  Scored from 1 to 5 where higher scores indicate increased appropriateness.
Feasibility of Intervention Measure (FIM) | post-test (up to 4 weeks)
  Scored from 1 to 5 where higher scores indicate increased feasibility.
HMP App Usage: Did you use the Healthy Minds Program App (Yes or No) | post-test (up to 4 weeks)
HMP App Usage: Did you download the Healthy Minds Program App (Yes or No) | post-test (up to 4 weeks)

SECONDARY OUTCOMES:
Change in Perceived Stress Score | baseline and post-test (up to 4 weeks)
  A measure of perceived stress in the past week scored from 0 to 4 where higher numbers indicate higher stress.
Change in WHO-5 Well-Being Score | baseline and post-test (up to 4 weeks)
  A measure of well-being in the past week scored from 1 to 6 where higher numbers indicate greater well-being.
Change in PROMIS Depression Score | baseline and post-test (up to 4 weeks)
  A measure of feelings of depression scored from 1 to 5 where higher numbers indicate increased feelings of depression.
Change in PROMIS Anxiety Score | baseline and post-test (up to 4 weeks)
  A measure of feelings of anxiety scored from 1 to 5 where higher numbers indicate increased feelings of anxiety.
Change in Meaning of Life Questionnaire - Presence Subscale Score | baseline and post-test (up to 4 weeks)
  Scored from 1 to 7 where higher scores indicate greater sense of meaning and purpose.
Change in NIH Toolbox Loneliness Score | baseline and post-test (up to 4 weeks)
  A measure of loneliness scored from 1 to 5 where higher scores indicate increased loneliness.
Change in Suicide Cognitions Scale Score | baseline and post-test (up to 4 weeks)
  A 16-item survey scored from 0-4 for a total range of scores from 0-64. Higher scores indicate increased suicidal cognition.
HMP App Usage: How many times did you use the HMP App | post-test (up to 4 weeks)
  Tally of participant usage from 1 time, less than once per week, about once per week, more than once per week, about daily.

OTHER OUTCOMES:
HMP App Usage: Reasons for not downloading the HMP App | post-test (up to 4 weeks)
  Tally of participant reasons, including not interested, not relevant, worried about data security, did not have time, or other.
HMP App Usage: Reasons for not opening the HMP App | post-test (up to 4 weeks)
  Tally of participant reasons, including not interested, not relevant, worried about data security, did not have time, or other.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No